CLINICAL TRIAL: NCT06388525
Title: Post-ERCP Cholecystectomy. How ERCP and ERCP-related Variables Effect the Outcomes?
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasir Musa Kesgin, MD, MD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: PostERCPLC
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography; ERCP-Laparoscopic Cholecystectomy Interval; Number of Preoperative ERCPs; Stone Extraction Status in ERCP Procedures; Biliary Stents; Mechanical Lithotripsy
Keywords: Endoscopic Retrograde Cholangiopancreatography; Laparoscopic Cholecystectomy; Subtotal Cholecystectomy
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERCP Group: All patients aged 18 years and over who underwent elective cholecystectomy surgery after a prior ERCP with a diagnosis of symptomatic cholelithiasis and whose surgery was started laparoscopically
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography
- Standard/Non-ERCP Group: All patients aged 18 years and over who underwent elective cholecystectomy surgery without an ERCP history with a diagnosis of symptomatic cholelithiasis and whose surgery was started laparoscopically

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreatography
  Groups: ERCP Group

SUMMARY:
In this retrospective study, we aimed to detect of effects of ERCP on outcomes of Laparoscopic Cholecystectomy. Patients underwent elective cholecystectomy surgery with a diagnosis of symptomatic cholelithiasis were identified and divided into two main groups regarding to have a ERCP procedure prior to surgery or not. To eliminate possible differences in baseline characteristics, patients in ERCP and non-ERCP groups were propensity score-matched 1:1 using nearest-neighbor matching without replacement based on age, sex and ASA score. Following propensity score matching (PSM), the ERCP and non-ERCP groups were first compared to detect effects of the ERCP procedure itself. After comparison of two main groups, subgroup analyzes performed for the ERCP group to detect effect of ERCP-related variables (indication for ERCP procedure, time between last ERCP procedure and surgery, number of preoperative ERCPs, stone extractions, and biliary stent use)

DETAILED DESCRIPTION:
All patients aged 18 years and over who underwent elective cholecystectomy surgery with a diagnosis of symptomatic cholelithiasis and whose surgery was started laparoscopically in a single tertiary reference hospital between January 1, 2016 and January 1, 2020 were identified retrospectively using the hospital data. Patients with a diagnosis of malignancy, with a history of percutaneous cholecystostomy, who underwent cholecystectomy while being operated for a different indication, and those who were diagnosed with cholecystoenteric fistula during the operation, were excluded from the study. After exclusion, patients first divided to two groups regarding to have a ERCP procedure prior to surgery or not. Age, sex, ASA scores, history of previous abdominal surgery, Charlson Comorbidity Index (CCI) values were included as baseline data. In terms of CCI scores, patients categorized into two subgroups according to CCI scores greater than 3 or not. To eliminate possible differences in baseline characteristics, patients were propensity score-matched 1:1 using nearest-neighbor matching without replacement based on age, sex and American Society of Anesthesiologists (ASA) score. Following propensity score matching (PSM), the ERCP and non-ERCP groups were first compared to detect effects of the ERCP procedure itself.

The primary outcomes examined in our study were conversion to open and subtotal cholecystectomy, intraoperative adhesion levels and operative time, hospital stay and postoperative complications. Only complications that have a Clavien-Dindo Score greater or equal to 3 were noted as postoperative complication for analyzes. While the patients with no adhesions were considered as group A, the patients with adhesions covering less than 50% of the gallbladder were considered as group B, whereas the patients in whom the gallbladder was completely covered with adhesions were considered as group C.

After comparison of two main groups, subgroup analyzes performed for the ERCP group to detect effect of ERCP-related variables to the same outcomes. The variables used in each separate subgroup analysis in the ERCP group were as follows: indication for ERCP procedure, time between last ERCP procedure and surgery, number of preoperative ERCPs, stone extractions, and biliary stent use. Information about mechanical lithotripsy was also noted and used for a separate subgroup analysis

For the first subgroups analysis, ERCP group divided into two subgroups regarding the preoperative ERCP indication was cholangitis or not. The second subgroup analysis was based on the ERCP-Laparoscopic cholecystectomy interval and three subgroups determined. Accordingly, for the timing of surgery, the first two weeks after ERCP were classified as early interval, the 2nd and 6th weeks as moderate interval, and the 6 weeks or later after ERCP, as late interval. Each of the number of preoperative ERCPs, extracted stones, and placed biliary stents were also used determinants for shaping the other subgroups. For the design of the last subgroup, patients were divided into two subgroups according to whether or not they had mechanical lithotripsy in their preoperative ERCP.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and over who underwent elective cholecystectomy surgery with a diagnosis of symptomatic cholelithiasis and whose surgery was started laparoscopically

Exclusion Criteria:

* Patients with a diagnosis of malignancy, with a history of percutaneous cholecystostomy, who underwent cholecystectomy while being operated for a different indication, and those who were diagnosed with cholecystoenteric fistula during the operation, were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After exclusion, patients first divided to two groups regarding to have a ERCP procedure prior to surgery or not. Age, sex, ASA scores, history of previous abdominal surgery, Charlson Comorbidity Index (CCI) values were included as baseline data. In terms of CCI scores, patients categorized into two subgroups according to CCI scores greater than 3 or not. To eliminate possible differences in baseline characteristics, patients were propensity score-matched 1:1 using nearest-neighbor matching without replacement based on age, sex and American Society of Anesthesiologists (ASA) score. Following propensity score matching (PSM), the ERCP and non-ERCP groups were first compared to detect effects of the ERCP procedure itself.
Sampling Method: Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Conversion to open | 2016-2020
  Decision to continue with conventional open surgery despite laparoscopic initiation
Subtotal Cholecystectomy | 2016-2020
  Decision to complete the procedure with a subtotal cholecystectomy, despite an initial goal of a total cholecystectomy
Postoperative Complications | 2016-2020
  Any postoperative complications that have a Clavien-Dindo Score greater than or equal to 3
Adhesion levels | 2016-2020
  Perivesical adhesion status based on descriptions of omental adhesion levels defined by Sugrue et al.
Operative time | 2016-2020
  Duration of surgical procedure itself
Length of hospital stay | 2016-2020
  Time spent in hospital until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Musa Kesgin, Principal Investigator — Istanbul Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The participant data are not publicly available due to institutional policies but are available from the corresponding author on reasonable request